CLINICAL TRIAL: NCT02554578
Title: Effectiveness Improving Medication Adherence in Heart Transplant Management
Brief Title: Impact of mHealth in Heart Transplant Management
Acronym: mHeart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-MHE-2014-55
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Heart Transplant
Keywords: mHealth; multidisciplinary team; immunosuppressive medication; pharmaceutical care; adherence; heart transplant; recipients
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmaceutical care programme supported by mHealth (Experimental)
  Interventions: Other: Multidisciplinary follow-up programme supported by mHealth
- Routine healthcare by the transplant team (No Intervention)

INTERVENTIONS:
Other: Multidisciplinary follow-up programme supported by mHealth — The follow-up programme integrates an online health platform (app and web) to monitor patients remotely, into the multidisciplinary team workflow, in order to improve heart transplant management.
  Patients will use the mobile application designed to help them to manage their health issues and facilitate communication with the transplant team.
  Data recorded manually by the patient using the mHealth application include pharmacotherapeutic information (medication adherence, barriers to adherence, side effects, interactions, etc.), clinical symptoms and other relevant clinical information (blood pressure, cardiac frequency, exercise, glucose level, diet, mood, etc.).
  mHealth will be used by the transplant team as a complementary way of deliver patient care. Analysis of the data collected by the multidisciplinary team may help to prioritise and provide personalized pharmacotherapeutic and medical interventions to patients and their families.
  Other Names: Heart transplantation management by a multidisciplinary team and supported by mobile health (mHealth)
  Arms: Pharmaceutical care programme supported by mHealth

SUMMARY:
The purpose of this study is to improve medication adherence, engagement and support to heart transplant patients through implementation of a new clinical care programme conducted by the clinical pharmacy service in cooperation with the heart transplant team and supported by mobile health (mHealth).

DETAILED DESCRIPTION:
Non-adherence to immunosuppressive medications generally ranges from 20-40% and is associated with acute rejection episodes and graft loss. Many solid organ transplant centres have incorporated transplant pharmacists into the multidisciplinary transplant clinical team focused on improving outcomes and safety associated with drug therapy.

Mobile technology has undergone rapid advances in the past several years and the use of mHealth in pharmaceutical care is changing pharmacy practice. Several published reports have identified general mobile applications suited for improve adherence. But evidence supporting the benefits in clinical practice is limited.

This study expects to analyse the potential of mHealth to improve medication adherence and heart transplant patient management in real clinical practice.

The investigators asses a new multidisciplinary follow-up programme in heart transplant recipients supported by mobile health (mHealth) with the aim to improve medication adherence, prevent drug related problems and improve patient clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant patients ≥ 18 years of age
* Give informed consent.
* Be able to use a mobile device (smartphone).
* Sign a confidentiality agreement (interventional group).

Exclusion Criteria:

* Do not meet all the inclusion criteria.
* Non-available to receive a minimum of one-year clinical follow-up by the heart transplant unit.
* Suffer severe mental disorders, other mental pathologies or conditions that can be a barrier to use the mobile application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Medication adherence measured on validated scales and questionnaires | 6 months
  Change From Baseline in Medication Adherence on the Simplified Medication Adherence Questionnaire (SMAQ)

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829